CLINICAL TRIAL: NCT02857517
Title: Intravitreal Conbercept for Idiopathic Choroidal Neovascularization
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiao Mingfei (Other)
Responsible Party: Sponsor-Investigator, Jiao Mingfei, Principal Investigator, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJMUEH001
Record Dates: First submitted 2016-07-27; First posted 2016-08-05 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Idiopathic Choroidal Neovascularization
MeSH Terms: interventions — KH902 fusion protein

ARMS (1):
- intravitreal 0.05ml conbercept for ICNV (Experimental): 0.05ml conbercept ,1 injection with PRN
  Interventions: Drug: conbercept

INTERVENTIONS:
Drug: conbercept — 0.05ml conbercept
  Other Names: conbercept fusion protein

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravitreal anti-vascular endothelial growth factor (anti-VEGF) therapy as primary treatment for ICNV.

ELIGIBILITY:
Inclusion Criteria:

* Patient who give voluntary signed informed consent
* Patient affiliated with the Tianjin Medical University Eye Hospital or similar
* Patient with ICNV with active primary subfoveal, retrofoveal or juxtafoveal lesions that affect the fovea as evidenced by angiography (fluorescein and/or indocyanin green) and/or SD-OCT in the studied eye
* Patient willing, committed and able to return for all clinic visits and complete all study-related procedures

Exclusion Criteria:

* Pregnant women
* Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study
* Patient who is protected adults according to the terms of the law (French public health laws)
* Involvement in another clinical trial (studied eye and/or the other eye)
* Patient with non-ICNV, especially:

  * AMD
  * High myopia defined as refraction ≥ - 6 diopters
* Other curative treatment of ICNV in the studied eye during the last 3 months before the first intravitreal injection: anti-VEGF therapy, juxta- or extra-foveal macular laser, photodynamic therapy, surgery, external radiotherapy, transpupillary thermotherapy ...
* Medical history of retrofoveal focal macular laser photocoagulation in the studied eye
* Subretinal haemorrhage reaching the fovea centre, with a size > 50% of the lesion area
* Fibrosis or retrofoveal retinal atrophy in the studied eye
* Retinal pigment epithelial tear reaching the macula in the studied eye
* Medical history of intravitreal medical device in the studied eye
* Medical history of auto-immune or idiopathic uveitis
* Proved diabetic retinopathy
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments
* Aphakia or lack of lens capsule (not removed by YAG laser) in the studied eye
* Arterial hypertension that is not controlled by an appropriate treatment
* Previous or actual treatment with systemic administration of anti-VEGF therapy
* Known hypersensitivity to aflibercept, or another drug composite of the medicinal product used; allergy to fluorescein, indocyanin green, anaesthetic eye drops
* Active or suspected ocular or peri-ocular infection
* Serious active intra-ocular inflammation in the studied eye
* Medical history of intra-ocular surgery within 28 days before the first injection in the studied eye
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion
* Follow up not possible during 12 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
visual acuity(Snellen chart) | baseline
visual acuity(Snellen chart) | Change from Baseline visual acuity at one day after injection
visual acuity(Snellen chart) | Change from Baseline visual acuity at one week after injection
visual acuity(Snellen chart) | Change from Baseline visual acuity at four weeks after injection
visual acuity | Change from Baseline visual acuity at eight weeks after injection
visual acuity(Snellen chart) | Change from Baseline visual acuity at 12weeks after injection
visual acuity(Snellen chart) | Change from Baseline visual acuity at half year after injection
visual acuity(Snellen chart) | Change from Baseline visual acuity at 1 year after injection

SECONDARY OUTCOMES:
macular central fovea thickness(OCT) | baseline
macular central fovea thickness | Change from Baseline macular central fovea thickness at four weeks after injection
macular central fovea thickness(OCT) | Change from Baseline macular central fovea thickness at eight weeks after injection
macular central fovea thickness(OCT) | Change from Baseline macular central fovea thickness at 12 weeks after injection
macular central fovea thickness(OCT) | Change from Baseline macular central fovea thickness at half year after injection
macular central fovea thickness(OCT) | Change from Baseline macular central fovea thickness at 1 year after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China